CLINICAL TRIAL: NCT01908244
Title: Short-term Effects of Live Pentatonic Music on Physiological Parameters in Preterm Infants - A Randomized Controlled Trial With Crossover Design
Brief Title: Short-term Effects of Live Music in Preterm Infants
Acronym: MTN05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ARCIM_MTN05
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-07

CONDITIONS: Prematurity
Keywords: Preterm infants, music, Neonatal Intensive Care Unit (NICU)
MeSH Terms: conditions — Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Control (No Intervention): No pentatonic music
- Music (Experimental)
  Interventions: Other: Music

INTERVENTIONS:
Other: Music — Pentatonic music
  Arms: Music

SUMMARY:
The purpose of this study is to determine the effects of pentatonic live music on physiological parameters in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 26-34 weeks; no use of CPAP (Continous Positive Airway Pressure) or any other form of mechanical ventilation; signed informed consent of the parents

Exclusion Criteria:

* Heart defect or known cardiac arrhythmia; other diseases of the preterm and newborn period (including infections and chromosomal aberrations) which make an additional diagnostic and therapeutic intervention unacceptable; detection of deafness (TEOAE, transitory evoked otoacoustic emission)

Ages: 26 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Numbers of desaturations < 90% per hour | physiological parameters are measured twice over a period of 2 hours and 15 minutes

SECONDARY OUTCOMES:
DI < 85% (Desaturations <85%/hour) | Physiological parameters are measured twice over a period of 2 hours and 15 minutes.
DI < 80% (Desaturations <80% per hour) | Physiological parameters are measured twice over a period of 2 hours and 15 minutes.
Heart rate | Physiological parameters are measured twice over a period of 2 hours and 15 minutes.
Oxygen saturation | Physiological parameters are measured twice over a period of 2 hours and 15 minutes.
Apnoea > 4 sec /h | Physiological parameters are measured twice over a period of 2 hours and 15 minutes.
Bradycardia < 80 bpm/h | Physiological parameters are measured twice over a period of 2 hours and 15 minutes.
Tachycardia > 200 bmp/h | Physiological parameters are measured twice over a period of 2 hours and 15 minutes.
HRV-Parameters | Physiological parameters are measured twice over a period of 2 hours and 15 minutes.
  SDNN, RMSSD, pNN50, LF/HF
PI | Physiological parameters are measured twice over a period of 2 hours and 15 minutes.
  Perfusionindex
PTT | Physiological parameters are measured twice over a period of 2 hours and 15 minutes.
  Pulse-Transit-Time (ms)
State Trait Anxiety Inventory | If present questionnaires are filled in by the child's mother before and after the music intervention respectively no intervention
State of the child | If present questionnaires are filled in by the child's mother before and after the music intervention respectively no intervention
additional music questions | If present questionnaires are filled in by the child's mother before and after the music intervention respectively no intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Filderklinik, Filderstadt, Baden-Wurttemberg
  - Universtitätsklinikum für Kinder und Jugendmedizin, Abteilung IV Neonatologie, Tübingen, Baden-Wurttemberg

REFERENCES:
- [Background] Arnon S, Shapsa A, Forman L, Regev R, Bauer S, Litmanovitz I, Dolfin T. Live music is beneficial to preterm infants in the neonatal intensive care unit environment. Birth. 2006 Jun;33(2):131-6. doi: 10.1111/j.0730-7659.2006.00090.x. PMID 16732778
- [Background] Standley JM. A meta-analysis of the efficacy of music therapy for premature infants. J Pediatr Nurs. 2002 Apr;17(2):107-13. doi: 10.1053/jpdn.2002.124128. PMID 12029604